CLINICAL TRIAL: NCT01694108
Title: Bacille Calmette Guérin Immunisation at Birth and Childhood Morbidity in Danish Children. A Prospective, Randomised, Clinical Trial.
Brief Title: Bacille Calmette Guérin Immunisation at Birth and Childhood Morbidity in Danish Children.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lone Graff Stensballe (Other)
Collaborators: Hvidovre University Hospital (Other); Kolding Sygehus (Other); Danish National Research Foundation (Other); Research Center for Vitamins and Vaccines (CVIVA) (Unknown)
Responsible Party: Sponsor-Investigator, Lone Graff Stensballe, MD, PhD, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: EudraCT2010-021979-85
Record Dates: First submitted 2012-09-22; First posted 2012-09-26 (Estimated); Results first posted 2016-01-08 (Estimated); Last update posted 2017-05-24 (Actual); Status verified 2017-04

CONDITIONS: Prospective; Single-blind; Clinical; Trial; Intervention
MeSH Terms: interventions — BCG Vaccine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BCG-vaccine (SSI) (Experimental): Children born to mothers, who have accepted to participate, will be randomised to either intervention group or to the control group at birth. Block-randomisation stratified by hospital, gender and gestational age (≥37 weeks of gestation vs. < 37 weeks of gestation) will be performed electronically just before vaccination by the overall study electronic case report system (e-crf).
  Children randomised to the BCG vaccination group will receive an intradermal BCG vaccine (Statens Serum Institute "CG vaccine" in the standard dose 0.05 ml in the upper, lateral part of the arm of the child by a specially trained midwife or a study physician.
  Interventions: Biological: BCG-vaccine (SSI)
- No Intervention (No Intervention): Control children will be treated as usual, since no suitable placebo exists.

INTERVENTIONS:
Biological: BCG-vaccine (SSI)
  Arms: BCG-vaccine (SSI)

SUMMARY:
In high-income societies the use of health care and medication is steadily increasing. Children have high morbidity, many visits at the general practitioner, an increasing number of hospitalisations, and an increasing use of medication. And, when children are ill, someone has to stay home to care for them. An un-explained global increase in the incidence of the allergic diseases eczema, wheezing, asthma and allergies means that 25% of high-income populations are affected. Cheap preventive measures are highly warranted. Recent studies have shown a positive, non-specific effect of early Bacille Calmette Guérin (BCG) immunisation on neonatal mortality in low-income countries and suggested a positive, non-specific effect on allergic disease in high-income countries. "Non-specific" means that the vaccine effect goes beyond prevention of the targeted disease, i.e. the BCG vaccine benefits the health status of the immunised individual in ways unrelated to protection against tuberculosis (TB). For instance, in a recent randomised trial in West Africa the investigators showed that the BCG vaccine at birth was safe in low birth weight (LBW) infants and significantly reduced neonatal mortality in these children, with a significant long-lasting effect on infant mortality in the smallest newborns with a birth weight <1.5 kg. There is an urgent need to explore the huge potential of the BCG's beneficial immune-stimulatory effects among children in high-income populations.

Therefore, the investigators will carry out a large prospective randomised clinical trial in Denmark primarily designed to test the hypothesis that infants who get the BCG vaccine at birth experience 20% fewer hospitalisations during early childhood.

Secondary outcomes

1. To test the hypothesis that infants who get the BCG vaccine at birth are prescribed less antibiotics during early childhood than non-BCG-immunised infants.
2. To test the hypothesis that Danish infants who get the BCG vaccine at birth develop less eczema, asthmatic bronchitis/wheeze and food allergy at 3 and 12 months of age: self-reported, diagnosed by a physician, or found at clinical examination; and are prescribed less anti-eczema/asthma/allergy medication during early childhood than non-BCG-immunised infants.
3. To test the hypothesis that infants who receive the BCG at birth respond in paraclinical measures: Specific IgE, thymic gland size, leucocyte count and differentiation, monocyte memory, cytokine profiles, and antibody titres following immunisation against diphtheria, tetanus, pertussis, pneumococcus, hemophilus.
4. To test the hypothesis that infants who get the BCG vaccine at birth respond in growth measures: weight, length and head circumference.
5. To test the hypothesis that infants who get the BCG vaccine at birth respond with decreased morbidity: common cold, pneumonia, febrile episodes, diarrhoea and vomiting, acute otitis media, febrile convulsions.
6. To test the hypothesis that premature infants with gestational age less than 37 weeks who get the BCG vaccine at birth have unaffected psychomotor development measures: Ages and Stages scores.
7. To test the hypothesis that infants who get the BCG vaccine at birth has unaffected coverage with the subsequent vaccinations in the Child Vaccination Programme.
8. To test the above mentioned hypotheses specifically in the strata of premature and low-birth-weight Danish infants.

ELIGIBILITY:
Inclusion Criteria:

* All parents planning to give birth at Rigshospitalet, Hvidovre Hospital and Kolding Hospital will receive at letter during 2nd/3rd trimester of pregnancy with information on the study and be offered inclusion in the study.

Exclusion Criteria:

* Infants born before gestational age 32 weeks and/or birth weight < 1000g, infants with known congenital disease, anomaly or malformation, immune deficiency and HIV, will be excluded. Non-Danish speaking parents will be excluded.

Max Age: 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4262 (Actual)
Dates: Start 2012-09; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lone G Stensballe, MD, PhD, Principal Investigator — Rigshospitalet. The Danish National Hospital in Denmark.
Locations (3):
- Denmark (3):
  - Rigshospitalet, Copenhagen, Copenhagen Ø
  - Hvidovre Hospital, Copenhagen
  - Kolding Sygehus, Kolding

REFERENCES:
- [Derived] Dybdal D, Stensballe LG, Greisen G, Kjaergaard J. Validity of parent-reported weight and length of infants. Dan Med J. 2023 Aug 23;70(9):A11220712. PMID 37622649
- [Derived] Birk NM, Nissen TN, Ladekarl M, Zingmark V, Kjaergaard J, Jensen TM, Jensen SK, Thostesen LM, Kofoed PE, Stensballe LG, Andersen A, Pryds O, Nielsen SD, Benn CS, Jeppesen DL. The association between Bacillus Calmette-Guerin vaccination (1331 SSI) skin reaction and subsequent scar development in infants. BMC Infect Dis. 2017 Aug 3;17(1):540. doi: 10.1186/s12879-017-2641-0. PMID 28774269
- [Derived] Stensballe LG, Sorup S, Aaby P, Benn CS, Greisen G, Jeppesen DL, Birk NM, Kjaergaard J, Nissen TN, Pihl GT, Thostesen LM, Kofoed PE, Pryds O, Ravn H. BCG vaccination at birth and early childhood hospitalisation: a randomised clinical multicentre trial. Arch Dis Child. 2017 Mar;102(3):224-231. doi: 10.1136/archdischild-2016-310760. Epub 2016 Jul 21. PMID 27443836
- [Derived] Kjaergaard J, Birk NM, Nissen TN, Thostesen LM, Pihl GT, Benn CS, Jeppesen DL, Pryds O, Kofoed PE, Aaby P, Greisen G, Stensballe LG. Nonspecific effect of BCG vaccination at birth on early childhood infections: a randomized, clinical multicenter trial. Pediatr Res. 2016 Nov;80(5):681-685. doi: 10.1038/pr.2016.142. Epub 2016 Jul 18. PMID 27429204
- [Derived] Kjaergaard J, Stensballe LG, Birk NM, Nissen TN, Thostesen LM, Pihl GT, Nielsen AV, Kofoed PE, Aaby P, Pryds O, Greisen G. Bacillus Calmette-Guerin vaccination at birth: Effects on infant growth. A randomized clinical trial. Early Hum Dev. 2016 Sep;100:49-54. doi: 10.1016/j.earlhumdev.2016.05.015. Epub 2016 Jul 7. PMID 27394195
- [Derived] Kjaergaard J, Stensballe LG, Birk NM, Nissen TN, Foss KT, Thostesen LM, Pihl GT, Andersen A, Kofoed PE, Pryds O, Greisen G. Lack of a Negative Effect of BCG-Vaccination on Child Psychomotor Development: Results from the Danish Calmette Study - A Randomised Clinical Trial. PLoS One. 2016 Apr 28;11(4):e0154541. doi: 10.1371/journal.pone.0154541. eCollection 2016. PMID 27123570
- [Derived] Nissen TN, Birk NM, Kjaergaard J, Thostesen LM, Pihl GT, Hoffmann T, Jeppesen DL, Kofoed PE, Greisen G, Benn CS, Aaby P, Pryds O, Stensballe LG. Adverse reactions to the Bacillus Calmette-Guerin (BCG) vaccine in new-born infants-an evaluation of the Danish strain 1331 SSI in a randomized clinical trial. Vaccine. 2016 May 11;34(22):2477-82. doi: 10.1016/j.vaccine.2016.03.100. Epub 2016 Apr 7. PMID 27060379

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BCG-vaccine | Control Children (no Intervention)
Started | 2129 | 2133
Completed | 2129 (100% follow-up) | 2133 (100% follow-up)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics by allocation among the 4184 mothers in The Danish Calmette Study
Groups:
- BCG-vaccine: SSI strain 1331 standard dose
- Control Children: No intervention
- Total: Total of all reporting groups
Arm/Group | BCG-vaccine | Control Children | Total
Number analyzed (Participants) | 2095 | 2089 | 4184
Age, Continuous [Mean (Standard Deviation); unit: years] — Maternal age
  years | 32.0 (4.6) | 31.9 (4.4) | 31.95 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender of the child. In multiple births: gender of the first born child.
  Participants
    Female | 1003 | 985 | 1988
    Male | 1092 | 1104 | 2196
Region of Enrollment [Number; unit: participants] — All three study sites are situated in Denmark.
  participants
    Denmark | 2095 | 2089 | 4184
Premature birth [Number; unit: participants] | 61 | 60 | 121

OUTCOME MEASURES:

1. Primary Outcome: All-cause Hospitalisations
Description: To test that infants who get the BCG vaccine at birth experience 20% fewer hospitalisations in early childhood than non-BCG-immunised infants.
Time Frame: 0-15 months of age
Population: Intention-to-treat
Measure: Number; unit: Events
Arm/Group | BCG-vaccine | Control Children (no Intervention)
Number analyzed (Participants) | 2129 | 2133
Events | 637 | 633

2. Secondary Outcome: Antibiotics
Description: To test that infants who get the BCG vaccine at birth are prescribed less antibiotics during early childhood than non-BCG-immunised infants. Use of antibiotics was defined as one or more precriptions of systemic antibiotics (ATC groups J01, J02, J05, all subgroups inclusive).
Time Frame: 0-15 months of age
Population: Intention-to-treat
Measure: Number; unit: participants
Arm/Group | BCG-vaccine | Control Children
Number analyzed (Participants) | 2129 | 2133
participants | 934 | 931

3. Secondary Outcome: Atopic Dermatitis
Description: To test if BCG vaccination within 7 days after birth influence the risk of atopic dermatitis defined by clinical examination at 13 months of age using "scoring atopic dermatitis (SCORAD)" or by parental report of physician diagnosed atopic dermatitis in the telephone interview at 13 months of age.
Time Frame: 13 months of age
Population: This analysis includes children with follow-up data from clinical examination or telephone interview. As opposed to the register-based primary outcome, adherence to telephone-interview and clinical examination was slightly lower than 100%.
Measure: Number; unit: participants
Groups:
- BCG-vaccine: SS! strain 1331 standard dose
Arm/Group | BCG-vaccine | Control Children
Number analyzed (Participants) | 2052 | 1952
participants | 466 | 495

4. Secondary Outcome: Specific IgE
Description: Number of participants with specific IgE (Phadiatop Infant) above the clinical cut-of level of 0.35.
Time Frame: 13 months of age
Population: This analysis includes children who participated with blood samples for this sub-study regarding specific IgE.
Measure: Number; unit: participants
Arm/Group | BCG-vaccine | Control Children
Number analyzed (Participants) | 743 | 627
participants | 55 | 50

5. Secondary Outcome: Standardized Weight at 13 Months
Description: To test that infants who get the BCG vaccine at birth respond in weight.The Z-score indicates the number of standard deviations away from the mean weight-for-age of the WHO anthropometric reference population (http://www.who.int/childgrowth/standards/en/). A Z-score of 0 is equal to the mean. Negative numbers indicate values lower than the mean and positive numbers indicate values higher than the mean.
Time Frame: 13 months of age
Population: This analysis only includes children with available follow-up data from telephone interviews or clinical examinations. As opposed to the primary outcome, follow-up was lower than 100%.
Measure: Mean (Standard Deviation); unit: Weight z-score at 13 months
Arm/Group | BCG-vaccine | Control Children
Number analyzed (Participants) | 2052 | 1950
Weight z-score at 13 months | 0.58 (0.90) | 0.61 (0.94)

6. Secondary Outcome: Psychomotor Development in Premature Infants
Description: To test that premature infants with gestational age less than 37 weeks who get the BCG vaccine at birth have unaffected psychomotor development measures: ASQ: Ages and stages questionnaire - a parent reported questionnaire that measures child psychomotor development. Total range of ASQ score: 0 to 300 points. Higher scores indicate higher level of psychomotor development.
Time Frame: 13 months of age
Population: This analysis only includes children from a particular subgroup (premature children, N = 144), who had with available follow-up data. As opposed to the primary outcome, follow-up was lower than 100%.
Measure: Mean (Standard Deviation); unit: Score on ASQ scale
Arm/Group | BCG-vaccine | Control Children
Number analyzed (Participants) | 56 | 59
Score on ASQ scale | 141.8 (53) | 153.5 (53.5)

7. Secondary Outcome: DTaP-IPV-Hib Vaccination Coverage at 12 Months of Age
Description: To test that infants who get the BCG vaccine at birth has unaffected coverage with the subsequent 3rd diphtheria, tetanus, acellular pertussis, polio, Haemophilus influenzae type b (DTaP-IPV-Hib) vaccination scheduled to 12 months of age according to the Danish child vaccination programme. Since we did not expect all children to get their immunizations exactly at 12 months of age, the children were followed up until 13-months of age.
Time Frame: 13 months of age
Population: Per-protocol analysis excluding 11 children randomised to BCG who did not receive the vaccine, and 36 children randomised to control who received the BCG vaccine.
Measure: Number; unit: participants
Arm/Group | BCG-vaccine | Control Children
Number analyzed (Participants) | 2018 | 2097
participants | 1175 | 1207

8. Secondary Outcome: Standardized Weight, Length and Head Circumference of Premature Children at 13 Months
Description: The Z-score indicates the number of standard deviations away from the mean weight-for-age of the WHO anthropometric reference population (http://www.who.int/childgrowth/standards/en/). A Z-score of 0 is equal to the mean. Negative numbers indicate values lower than the mean and positive numbers indicate values higher than the mean.
Time Frame: 13 months of age
Population: Premature children born with gestational age 32-36 weeks. This analysis only includes children from a particular subgroup (premature children, N = 144), who had with available follow-up data. As opposed to the primary outcome, follow-up was lower than 100%.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | BCG-vaccine | Control Children
Number analyzed (Participants) | 63 | 61
z-score
  Weight | 0.33 (0.95) | 0.34 (1.03)
  Length | 0.10 (0.97) | 0.02 (1.00)
  Head circumference | 0.51 (0.97) | 0.57 (0.99)

9. Secondary Outcome: Episodic Viral Wheeze
Description: Number of participants diagnosed with episodic viral wheeze by a physician and treated with anti-asthmatic medicine according to the telephone interview.
Time Frame: 13 months
Population: This analysis only includes children with available follow-up telephone interview data. As opposed to the primary outcome, follow-up was lower than 100%.
Measure: Number; unit: participants
Arm/Group | BCG-vaccine | Control Children
Number analyzed (Participants) | 2108 | 2081
participants | 211 | 195

10. Secondary Outcome: Food Allergy
Description: Number of participants with food allergy diagnosed by a physician and mentioned in the telephone interview at 13 months of age
Time Frame: 13 months
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | BCG-vaccine | Control Children
Number analyzed (Participants) | 2107 | 2076
participants | 15 | 10

11. Secondary Outcome: Length at 13 Months of Age
Description: To test if infants who get the BCG vaccine at birth respond in length. The Z-score indicates the number of standard deviations away from the mean weight-for-age of the WHO anthropometric reference population (http://www.who.int/childgrowth/standards/en/). A Z-score of 0 is equal to the mean. Negative numbers indicate values lower than the mean and positive numbers indicate values higher than the mean.
Time Frame: 13months
Population: This analysis only includes children with available follow-up data. As opposed to the primary outcome, follow-up for this outcome was lower than 100%.
Measure: Mean (Standard Deviation); unit: Length z-score
Arm/Group | BCG-vaccine | Control Children
Number analyzed (Participants) | 2050 | 1947
Length z-score | 0.54 (0.99) | 0.55 (1.00)

12. Secondary Outcome: Standardized Head Circumference at 13 Months of Age
Description: To test if infants who get the BCG vaccine at birth respond in head circumference. The Z-score indicates the number of standard deviations away from the mean weight-for-age of the WHO anthropometric reference population (http://www.who.int/childgrowth/standards/en/). A Z-score of 0 is equal to the mean. Negative numbers indicate values lower than the mean and positive numbers indicate values higher than the mean.
Time Frame: 13 months
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Head circumference z-score
Arm/Group | BCG-vaccine | Control Children
Number analyzed (Participants) | 2052 | 1952
Head circumference z-score | 0.78 (0.93) | 0.76 (0.95)

13. Secondary Outcome: Thymic Gland Size at 3 Months of Age
Description: To test that infants who receive the BCG at birth respond in thymic gland size defined by ultra sound examination. First, the thymus gland was identified in a horizontal scanning plane and the largest transverse diameter of the thymus was obtained. Second, in a sagittal scanning plane, the area of the largest lobe was assessed. Both measurements were obtained twice, and in case of more than 15% difference, both measurements were repeated. The mean of the two measurements were multiplied and defined as the thymic index.
Time Frame: 3 months of age
Population: This outcome was a sub-study to The Danish Calmette Study with 301 (BCG 153, Control 148) participating children.
Measure: Mean (95% Confidence Interval); unit: Thymic index
Arm/Group | BCG-vaccine | Control Children
Number analyzed (Participants) | 153 | 148
Thymic index | 33.10 [31.22 to 34.81] | 34.24 [32.42 to 36.16]

14. Secondary Outcome: Leucocyte Count 4 Days After Randomisation/Vaccination
Description: To test if infants who receive the BCG at birth respond in leucocyte count (white blood cell count) measured as geometric mean (GM) cell concentrations (GM*10^9 cells/L).
Time Frame: 4 days after randomisation/vaccination within 7 days after birth
Population: This was a sub study among 153 children with blood-samples at 4 days after randomisation/vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: cell concentrations (GM*10^9 cells/L)
Arm/Group | BCG-vaccine | Control Children
Number analyzed (Participants) | 75 | 78
cell concentrations (GM*10^9 cells/L) | 10.59 [10.06 to 11.15] | 10.70 [10.24 to 11.17]

15. Secondary Outcome: Monocyte Count 4 Days After Randomisation/Vaccination
Description: To test if infants who receive the BCG at birth respond in monocyte count measured as geometric mean (GM) cell concentrations (GM*10^9 cells/L).
Time Frame: 4 days after randomisation/vaccination within 7 days after birth
Population: This was a sub study among 153 children with blood-samples at 4 days after randomisation/vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: Cell concentrations (GM*10^9 cells/L)
Arm/Group | BCG-vaccine | Control Children
Number analyzed (Participants) | 75 | 78
Cell concentrations (GM*10^9 cells/L) | 1.58 [1.47 to 1.70] | 1.71 [1.60 to 1.82]

16. Secondary Outcome: Interferon Gamma Response
Description: To test that infants who receive the BCG at birth respond in interferon-gamma response upon stimulation with BCG. The interferon gamma response was defined as a value above the cut-off value of 107 pg/ml.
Time Frame: 13 months of age
Population: This is a sub study using bloodsamples. Only a small sub population from the overall trial participated.
Measure: Number; unit: participants
Arm/Group | BCG-vaccine | Control Children
Number analyzed (Participants) | 75 | 68
participants | 41 | 3

17. Secondary Outcome: Number of Participants With Antibody Concentration (AC) Against Tetanus of > 0.1 IU/mL
Description: To test the tetenus antibody response in BCG-vaccinated vs. non-BCG vaccinated children following routine immunisation against tetanus at 3, 5 and 12 months of age in blood samples obtained 13 months of age.
Time Frame: 13 months of age
Population: This outcome was a sub-study with 158 participants. Antibody concentration (AC) of > 0.1 IU/mL was considered protective
Measure: Number; unit: participants
Arm/Group | BCG-vaccine | Control Children
Number analyzed (Participants) | 80 | 78
participants | 80 | 78

18. Secondary Outcome: Number of Events of Common Cold
Description: To test that Danish infants who get the BCG vaccine at birth experience less events of common cold until 13 months of age than non-BCG-immunised infants.
Time Frame: 13 months of age
Population: as for outcome 11
Measure: Number; unit: Events
Arm/Group | BCG-vaccine | Control Children
Number analyzed (Participants) | 2096 | 2071
Events | 3990 | 3928

19. Secondary Outcome: Number of Events of Pneumonia
Description: To test that Danish infants who get the BCG vaccine at birth get less pneumonia at 13 months of age than non-BCG-immunised infants.
Time Frame: 13 months of age
Population: as for outcome 11
Measure: Number; unit: Events
Arm/Group | BCG-vaccine | Control Children
Number analyzed (Participants) | 2100 | 2070
Events | 207 | 162

20. Secondary Outcome: Number of Events of Febrile Episodes
Description: To test that Danish infants who get the BCG vaccine at birth get less febrile episodes at 13 months of age than non-BCG-immunised infants.
Time Frame: 13 months of age
Population: as for outcome 11
Measure: Number; unit: Events
Arm/Group | BCG-vaccine | Control Children
Number analyzed (Participants) | 2098 | 2069
Events | 1385 | 1302

21. Secondary Outcome: Number of Events With Diarrhoea and Vomiting
Description: To test that Danish infants who get the BCG vaccine at birth develop less episodes with diarrhoea and vomiting at 13 months of age than non-BCG-immunised infants.
Time Frame: 13 months of age
Population: as for outcome 11
Measure: Number; unit: Events
Arm/Group | BCG-vaccine | Control Children
Number analyzed (Participants) | 2103 | 2071
Events | 870 | 845

22. Secondary Outcome: Number of Events of Acute Otitis Media
Description: To test that Danish infants who get the BCG vaccine at birth develop less acute otitis media at 13 months of age than non-BCG-immunised infants.
Time Frame: 13 months of age
Population: as for outcome 11
Measure: Number; unit: Events
Arm/Group | BCG-vaccine | Control Children
Number analyzed (Participants) | 2098 | 2072
Events | 595 | 591

23. Secondary Outcome: Number of Events of Febrile Convulsions
Description: To test that Danish infants who get the BCG vaccine at birth develop less febrile convulsions at 13 months of age than non-BCG-immunised infants.
Time Frame: 13 months of age
Population: as for outcome 11
Measure: Number; unit: Events
Arm/Group | BCG-vaccine | Control Children
Number analyzed (Participants) | 2103 | 2070
Events | 44 | 25

24. Other Pre Specified Outcome: Decisional Conflict Scale Score
Description: After parents having made the decision about whether to accept vaccination of their newborn through participation in The Danish Calmette Study, O'Connor's Decisional Conflict Scale was used to identify decisional conflicts. The score ranges from 0 (no decisional conflict) til 100 (maximum decisional conflict). Scores lower than 25 are associated with implementing decisions; scores exceeding 37.5 are associated with decision delay or feeling unsure about implementation; so a low score reflects a low level of doubt about the decision about participation/decline participation in the trial, and a high score reflects a high level of doubt.
Time Frame: The decisional conflict score was measured before randomisation
Population: This outcome was a sub-study to The Danish Calmette Study with 667 participating mothers and 320 declining mothers.
Measure: Mean (Inter-Quartile Range); unit: decisional conflict score
Groups:
- Participating Mothers: Mothers who decided to let their child participate in the study
- Declining Mothers: Mothers who decided not to let their child participate in the study
Arm/Group | Participating Mothers | Declining Mothers
Number analyzed (Participants) | 667 | 320
decisional conflict score | 18.8 [0 to 53.1] | 17.2 [0 to 67.2]
Statistical Analysis 1: Comparison: Participating Mothers vs Declining Mothers; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney); Mann-Whitney-test comparing the decisional conflict scores of participating mothers vs. declining mothers

25. Other Pre Specified Outcome: Quality of Communication and Information
Description: To test that the use of telephone and internet was acceptable in the study population using the Quality of Informed Consent (QuIC) questionnaire. The questionnaire was divided into six categories; five on study comprehension and one on satisfaction with the information process. The items in the first five categories could be answered with "yes", "no" or "do not know". The last category was rated on a 7-point Likert scale, with 1 being "very dissatisfied" and 7 being "very satisfied". The primary outcome was the sum of the score for comprehension items and satisfaction items. Comprehension items were scored 1 point for each correct answer and 0 points for each incorrect answer. Satisfaction items were scored as rated on the 7-point Likert scale. Total score ranged from 7 to 69 points, comprehension score from 0 to 20 points and satisfaction score from 7 to 49 points. The higher score, the better comprehension and satisfaction.
Time Frame: 2 days after the information was given
Population: This is a small, separate sub-study. 59 + 59 participants had sufficient follow-up data to participate in the analysis.
Measure: Mean (Inter-Quartile Range); unit: Score on QuIC scale
Groups:
- Telephone: Randomized to receive information about the study by telephone
- Face-to-face: Randomized to receive information about the study by standard face-to-face consultation.
Arm/Group | Telephone | Face-to-face
Number analyzed (Participants) | 59 | 59
Score on QuIC scale | 61.40 [58 to 65] | 64.42 [63 to 67]

ADVERSE EVENTS:
Arm/Group | BCG-vaccine | Control Children (no Intervention)
Serious Adverse Events (participants affected / at risk) | 65/2129 | 45/2133
Other Adverse Events (participants affected / at risk) | 233/2129 | 123/2133
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BCG-vaccine (N=2129) | Control Children (no Intervention) (N=2133)
Dead (General disorders) | 3 (3) | 1 (1)
Other than dead (General disorders) | 62 (62) | 44 (44) — Registered as: life-threatening events, hospitalizations, events causing disability. No life-threatening events, or events causing disability were however registered.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BCG-vaccine (N=2129) | Control Children (no Intervention) (N=2133)
BCG-vaccine related event (Infections and infestations) | 212 (212) | 0 (0)
Other than BCG-vaccine related (General disorders) | 21 (2129) | 123 (2133)

LIMITATIONS AND CAVEATS:
The allocation was planned to be stratified by sex, study site, and prematurity, however, due to a programming error the allocation was stratified only by prematurity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No